CLINICAL TRIAL: NCT01900574
Title: A Phase 1b Open-Label Study to Assess the Safety and Pharmacokinetics of Subcutaneously Administered Golimumab, a Human Anti-TNFα Antibody, in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Subcutaneously Administered Golimumab, a Human Anti-TNFα Antibody, in Pediatric Patients With Moderate to Severe Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101676; CNTO148UCO1001 (Other: Janssen Research & Development, LLC); 2012-004366-18 (EudraCT Number)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; Ulcerative Colitis; Moderately to Severely Active Ulcerative Colitis; Golimumab; Simponi; Human anti-TNFα Antibody; Pediatric participants; Safety and Pharmacokinetics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Golimumab (Experimental)
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Golimumab will be administered subcutaneously. For participants weighing less than 45 kg, the dose of golimumab at Week 0 will be 90 mg/m2 (up to 200 mg) and 45 mg/m2 (up to 100 mg) at Weeks 2, 6, and 10. For participants weighing 45 kg or more, the dose of golimumab at Week 0 will be 200 mg and 100 mg at Weeks 2, 6, and 10. From Week 14, the dose of golimumab will be 45 mg/m2 and 100 mg, every 4 weeks for participants weighing less than 45 kg and 45 kg or more, respectively. From Week 18, participants weighing 45 kg or more have the option to administer golimumab at home after being properly trained. At Week 14 or at any time after, the participants have the option to decrease their dose of golimumab to 50 mg (weighing 45 kg or more) or 22.5 mg/square meter (less than 45 kg) at the discretion of the investigator. A single dose increase back to 100 mg or 45 mg/m2 is permitted based on the investigator's assessment of an increase in a participant's ulcerative colitis disease activity.
  Other Names: Simponi

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (what the body does to the study medication) and safety of subcutaneously (under the skin) administered golimumab in pediatric participants (aged 2 to 17 years) with moderately to severely active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
This is an open-label (both [participants and investigator] know what treatment participants will receive) and multicenter study. The study is divided into 2 parts: Part 1: pharmacokinetics portion (Week 0 to Week 14); Part 2: study extension (Week 14 to Week 114). The focus of this study is to evaluate the pharmacokinetics and safety of golimumab. Additionally the efficacy of short-term therapy with golimumab will be evaluated. Participants in clinical response at Week 6 will continue to receive open label golimumab maintenance therapy and will enter the study extension at Week 14. Participants who are not in clinical response at Week 6 will be withdrawn from further treatment with golimumab. At Week 114, participants who, in the opinion of the investigator, may benefit from continued treatment will be eligible to continue to receive golimumab every 4 weeks until marketing authorization is obtained in the treatment of pediatric UC in that country, or until a decision has been made not to pursue an indication in pediatric UC. Approximately 30 participants will be enrolled in this study. The total duration of study participation for a participant will be approximately 126 weeks or longer.

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe Ulcerative Colitis (UC) defined by a Mayo score (a score used to assess the treatment for UC) of 6 to 12 inclusive, including an endoscopic subscore of 2 or more.
* Must either be currently receiving treatment with, or have a history of having failed to respond to, or have a medical contraindication to at least 1 of the following therapies: oral or intravenous corticosteroids, 6-mercaptopurine and azathioprine OR must either have or have had a history of corticosteroid dependency (ie, an inability to successfully taper corticosteroids without a return of the symptoms of UC) OR required more than 3 courses of corticosteroids in the past year
* No history of latent or active tuberculosis prior to screening
* Positive protective antibody titers to varicella and measles prior to the first administration of study agent

Exclusion criteria:

* Have severe extensive UC that is likely to require a colectomy (surgical removal of the colon) within 12 weeks of study entry
* Have UC limited to the rectum only or to less than 20 cm of the colon
* Presence of a stoma
* Presence or history of a fistula
* Have evidence of Crohn's disease (an inflammatory large intestine disease)
* Previous exposure to anti-tumor necrosis factor therapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2015-02-18 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Serum golimumab concentrations at Week 6 | Week 6
  Sample will be collected prior to the administration of study medication.

SECONDARY OUTCOMES:
Number of participants who will achieve clinical response at Week 6 | Week 6
  Clinical response is defined as a decrease from baseline in the Mayo score by greater than or equal to 30 percent and greater than or equal to 3 points, with either a decrease from baseline in the rectal bleeding subscore of 1 or more or a rectal bleeding subscore of 0 or 1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe. Higher scores indicate worsening of the disease.
Number of participants who will achieve clinical remission at Week 6 measured by the Mayo score | Week 6
  Clinical remission is defined as a Mayo score less than or equal to 2 points, with no individual subscore greater than 1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe. Higher scores indicate worsening of the disease.
Number of participants who will achieve clinical remission at Week 6 measured by Pediatric Ulcerative Colitis Activity Index (PUCAI) score | Week 6
  Clinical remission is defined as a score less than 10 and it will be measured by the PUCAI scores, a noninvasive measure of ulcerative colitis disease activity. The PUCAI score consists of 6 scales (abdominal pain [points 0 to 10], rectal bleeding [points 0 to 30], stool consistency [points 0 to 10], number of stools [points 0 to 15], nocturnal bowel movement [points 0 to 10], and activity level [points 0 to 10]). The total score ranges from 0 and 85 points, where it is calculated as the sum of the 6 scales and decrease of 20 points is considered a minimally clinically important change. Higher scores indicates a more severe disease.
Number of participants with mucosal healing at Week 6 | Week 6
  Mucosal healing is calculated by endoscopy subscore of the Mayo score of 0 (normal or inactive disease) or 1 (mild disease).
Number of participants who will achieve clinical remission at Week 54 and Week 110 measured by Pediatric Ulcerative Colitis Activity Index (PUCAI) score | Week 54 and Week 110
  Clinical remission is defined as a score less than 10 and it will be measured by the PUCAI score, a noninvasive measure of ulcerative colitis disease activity. The PUCAI score consists of 6 scales (abdominal pain [points 0 to 10], rectal bleeding [points 0 to 30], stool consistency [points 0 to 10], number of stools [points 0 to 15], nocturnal bowel movement [points 0 to 10], and activity level [points 0 to 10]). The total score ranges from 0 and 85 points, where it is calculated as the sum of the 6 scales and decrease of 20 points is considered a minimally clinically important change. Higher scores indicates a more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- United States (9):
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Hartford, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Rochester, Minnesota
  - Morristown, New Jersey
  - Seattle, Washington
- Austria (2):
  - Graz
  - Vienna
- Brussels, Belgium
- Canada (3):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Toronto, Ontario
- Denmark (2):
  - Aarhus
  - Hvidovre
- Paris, France
- Germany (2):
  - Aachen
  - München
- Israel (3):
  - Beersheba
  - Haifa
  - Jerusalem
- Netherlands (2):
  - Nijmegen
  - Rotterdam
- Poland (2):
  - Rzeszow Poland
  - Warsaw